CLINICAL TRIAL: NCT06685120
Title: Combined Use of PRP and Hyaluronic Acid for Infiltrative Treatment of Patients With Knee Osteoarthritis - Randomized Controlled Clinical Study
Brief Title: Combined Use of PRP and Hyaluronic Acid for Infiltrative Treatment of Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP+HA-23
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee
Keywords: PRP; Platelet rich plasma; HA; Hyaluronic acid; PRP injection; PRP + HA injection; HA injection; Double-blind randomized controlled clinical trial

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomized controlled clinical trial with 1:1:1 allocation
Who Masked: Participant, Outcomes Assessor
Masking Description: They will be "blinded" patients, health care professionals who will assess clinical and functional outcomes (outcome assessors), and professionals who will analyze the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP+HA injection (Experimental): This group of patients randomized into the treatment group, will undergo single intra-articular injection of autologous PRP+HA
  Interventions: Combination Product: PRP + HA injection
- PRP injection (Active Comparator): This group of patients randomized into the treatment group, will undergo single intra-articular injection of autologous PRP
  Interventions: Biological: PRP injection
- HA injection (Active Comparator): This group of patients randomized into the treatment group, will undergo single intra-articular injection of HA
  Interventions: Device: HA injection

INTERVENTIONS:
Combination Product: PRP + HA injection — Following autologous PRP harvesting and production, 5 mL of PRP and 40 mg/2 mL of HA will be infiltrated into the knee joint affected by gonarthrosis. The combined procedure will be performed by first infiltrating the hyaluronic acid, and next, leaving the needle inserted into the joint to avoid a second needle insertion, the PRP will be infiltrated, respecting the conditions of sterility. In this way, the two products will not be mixed in the same syringe.
  Arms: PRP+HA injection
Biological: PRP injection — Following autologous PRP harvesting and production, patients randomized into control group 1 will undergo single intra-articular PRP infiltration. Five mL of PRP will be infiltrated into the knee joint affected by gonarthrosis.
  Arms: PRP injection
Device: HA injection — Patients randomized into control group 2, will undergo similar blood sampling as the PRP+ HA group and the PRP group to maintain blinding. They will then undergo intra-articular infiltration of 40 mg/ 2 ml HA into the knee with gonarthrosis.
  Arms: HA injection

SUMMARY:
"PRP+HA-23" is a double-blind randomized controlled clinical trial with 1:1:1 allocation. The objective of the study is to evaluate by a randomized controlled, double-blind clinical trial the efficacy and safety of viscosupplementation-associated PRP infiltration compared with PRP-only or HA-only infiltration for the treatment of patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Patients with osteoarthritis of the knee will be included in a randomized controlled, double-blind study, in which one group of patients will be treated with an infiltration of PRP combined with HA (PRP + HA group), one group of patients will be treated with an infiltration of PRP alone (PRP group), and another group of patients will be treated with an infiltration of HA alone (HA group). They will be "blinded" patients, health care professionals who will assess clinical and functional outcomes (outcome assessors), and professionals who will analyze the data.

A total of 288 patients will be included, and they will undergo infiltrative treatment after collecting informed consent for study participation and biographical data.

All enrolled patients undergo transfusion evaluation and venous whole blood sampling from 30 to 60 mL depending on the patient's hematocrit. From the withdrawn blood, which will be collected in tubes of 9 mL each, fresh autologous PRP (PRP) will subsequently be obtained. To maintain study blinding, all patients will have their blood drawn but PRP will not be produced for patients randomized into the HA group.Following autologous PRP harvesting and production, patients randomized into the treatment group will undergo single intra-articular infiltration of PRP + HA; patients randomized into the control group 1, will undergo single intra-articular infiltration of PRP; and patients randomized into the control group 2, will undergo similar blood sampling as the PRP+ HA group and the PRP group to maintain blindness. They will then undergo an intra-articular infiltration of HA .Patients will be clinically evaluated before the infiltration procedure and at 1-3-6- 12 and 24 months after treatment by medical personnel. Questionnaires will be administered for clinical evaluations before treatment and at the above-mentioned clinical checks during follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 40 to 75 years;
2. Patients with symptomatic knee osteoarthritis (VAS pain score between ≥ 3 and ≤ 8);
3. Unilateral involvement of symptomatology;
4. Radiographic or MRI signs of degenerative pathology of knee cartilage (Kellgren-Lawrence grade 1-3);
5. Failure, defined as the persistence of symptomatology, after at least one course of conservative treatment (pharmacological, physiotherapeutic or infiltrative treatment);
6. Hemoglobin > 11 g/dl; Platelet count > 150,000 plt/mm3 (Recently performed CBC examination);
7. Ability and consent of patients to actively participate in clinical follow-up;
8. Signature of informed consent.

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients undergoing intra-articular infiltration of other substance in the previous 6 months;
3. Patients undergoing knee surgery in the previous 12 months;
4. Patients with malignant neoplasms;
5. Patients with rheumatic diseases;
6. Patients with uncontrolled diabetes;
7. Patients with hematological diseases (coagulopathies);
8. Patients on anticoagulant-antiaggregant therapy that cannot be discontinued at the time of blood collection;
9. Patients with uncompensated thyroid metabolic disorders;
10. Patients abusing alcoholic beverages, drugs or medications;
11. Body Mass Index > 35;
12. Patients who have taken NSAIDs in the 3 days prior to blood draw;
13. Patients with cardiovascular disease for whom blood sampling 30 to 60 ml would be contraindicated;
14. Patients with recently performed CBC examination with Hb< 11 g/dl and Platelet values < 150,000 plt/mm3.
15. Pregnant and/or fertile women.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 1,3,6 and 24 months
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome
IKDC-Subjective Score (Subjective International Knee Documentation Committee) | baseline, 1,3,6, 12 and 24 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function.
  (Total score 0-100)
Objective parameters- Range of Motion | baseline, 1,3,6, 12 and 24 months
  Evaluation of the Range of Motion for comparative analysis.
Objective parameters - Circumferences | baseline, 1,3,6, 12 and 24 months
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis
Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline, 1,3,6, 12 and 24 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines the following categories: symptoms, stiffness, pain, daily activities, sports and quality of life.
  Each question is scored from 0 to 4, where 0 indicates "no difficulty" and 4 "severe difficulty. Score range 0-100 for each subscale
Visual Analogue Scale (VAS) (rest) | baseline, 1,3,6, 12 and 24 months
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" (0) and "the strongest pain imaginable" (10) during rest
Visual Analogue Scale (VAS) (exercise activity) | baseline, 1,3,6, 12 and 24 months
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" (0) and "the strongest pain imaginable" (10) during exercise activity
EuroQol Visual Analogue Scale (EQ-VAS) | baseline, 1,3,6, 12 and 24 months
  EQ-VAS is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
EQ-5D (EuroQoL) Current Health Assessment | baseline, 1,3,6, 12 and 24 months
  The generic health-related quality of life instrument-EQ-5D-allows both a description of health status along 5 dimensions and the evaluation of health or the estimation of a health summary score: the EQ-5D score on a scale where 0 is death and 1 is full health. EQ-5D is useful to evaluate the quality life of the patients. The EQ-5D respondents classify their own health status into 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with 3 levels of severity (no problems, moderate problems, or severe problems).
Tegner Activity Level Scale | baseline, 1,3,6, 12 and 24 months
  Tegner Activity Level Scale is a questionnaire to find out the patient's level of physical activity.All patients will indicate the type of sporting activity performed and its frequency.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability and 10 represents a competitive level of sport.
Patient Acceptable Symptom State (PASS) | baseline, 1,3,6, 12 and 24 months
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Final treatment opinion | 1,3,6, 12 and 24 months
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial. All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "", "much better", "somewhat better", "no change", "a little worse" ; "much worse"
Effectiveness of the blinding procedure | baseline
  The patient should indicate, after the infiltrative procedure, the type of treatment they think they received.The patient should choose from the following options:
  "PRP+HA infiltration," PRP infiltration", "HA infiltration". This question is designed to test the effectiveness of the blinding procedure
Expectations of treatment efficacy | baseline
  The patient should indicate at baseline what benefits they expect from the treatment.
  The patient should choose one of the following options:
  "Full recovery," "definitely better","much better", "somewhat better", "no change"

CONTACTS AND LOCATIONS:
Overall Officials: Davide Reale, MD, Principal Investigator — Istituto Ortopedico Rizzoli - Argenta
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Istituto Ortopedico Rizzoli, Bologna

REFERENCES:
- [Background] Boffa A, Salerno M, Merli G, De Girolamo L, Laver L, Magalon J, Sanchez M, Tischer T, Filardo G. Platelet-rich plasma injections induce disease-modifying effects in the treatment of osteoarthritis in animal models. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4100-4121. doi: 10.1007/s00167-021-06659-9. Epub 2021 Aug 2. PMID 34341845
- [Background] Filardo G, Previtali D, Napoli F, Candrian C, Zaffagnini S, Grassi A. PRP Injections for the Treatment of Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Trials. Cartilage. 2021 Dec;13(1_suppl):364S-375S. doi: 10.1177/1947603520931170. Epub 2020 Jun 19. PMID 32551947
- [Background] Chen WH, Lo WC, Hsu WC, Wei HJ, Liu HY, Lee CH, Tina Chen SY, Shieh YH, Williams DF, Deng WP. Synergistic anabolic actions of hyaluronic acid and platelet-rich plasma on cartilage regeneration in osteoarthritis therapy. Biomaterials. 2014 Dec;35(36):9599-607. doi: 10.1016/j.biomaterials.2014.07.058. Epub 2014 Aug 28. PMID 25176059
- [Background] Chiou CS, Wu CM, Dubey NK, Lo WC, Tsai FC, Tung TDX, Hung WC, Hsu WC, Chen WH, Deng WP. Mechanistic insight into hyaluronic acid and platelet-rich plasma-mediated anti-inflammatory and anti-apoptotic activities in osteoarthritic mice. Aging (Albany NY). 2018 Dec 23;10(12):4152-4165. doi: 10.18632/aging.101713. PMID 30582743
- [Background] Zhang Q, Liu T, Gu Y, Gao Y, Ni J. Efficacy and safety of platelet-rich plasma combined with hyaluronic acid versus platelet-rich plasma alone for knee osteoarthritis: a systematic review and meta-analysis. J Orthop Surg Res. 2022 Nov 19;17(1):499. doi: 10.1186/s13018-022-03398-6. PMID 36403041
- [Background] Lana JF, Weglein A, Sampson SE, Vicente EF, Huber SC, Souza CV, Ambach MA, Vincent H, Urban-Paffaro A, Onodera CM, Annichino-Bizzacchi JM, Santana MH, Belangero WD. Randomized controlled trial comparing hyaluronic acid, platelet-rich plasma and the combination of both in the treatment of mild and moderate osteoarthritis of the knee. J Stem Cells Regen Med. 2016 Nov 29;12(2):69-78. doi: 10.46582/jsrm.1202011. eCollection 2016. PMID 28096631